CLINICAL TRIAL: NCT02274129
Title: C51 - Clinical Survey of Oticon Medical Healing Cap
Brief Title: Clinical Survey of Oticon Medical Healing Cap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C51
Record Dates: First submitted 2014-10-14; First posted 2014-10-24 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Conductive Hearing Loss; Mixed Hearing Loss; Unilateral Partial Deafness
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Use of Healing cap II (Experimental): Single arm study using a new healing cap as intervention
  Interventions: Device: Healing cap II

INTERVENTIONS:
Device: Healing cap II — Healing cap II is used instead of the traditional healing cap as part of the surgical dressing after bone anchored hearing aid implant surgery

SUMMARY:
This study investigates the use of a new healing cap which, through altered design and choice of material, has been improved when it comes to minimizing the risk of it falling off as well as increasing patient comfort.

DETAILED DESCRIPTION:
This study will primarily investigate the use of a new healing cap, Healing cap II. The new healing cap has the same function as previous healing caps, but it soft instead of hard. Due to this, the healing cap is anticipated to not fall off as easily, but at the same time does not risk transferring larger forces than previously to the implant. Secondly, the patients will start using the sound processor 1-2 weeks after surgery. The implant stability will be monitored before and after loading by the use of resonance frequency analysis, an established method to evaluate and monitor osseointegrated implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for treatment with a bone anchored hearing aid
* 18 years or older

Exclusion Criteria:

* Inability to participate in follow-up
* Diseases or treatments known to compromise the bone quality at the implant site, e.g. radiotherapy, osteoporosis, diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-04-19 (Actual)

PRIMARY OUTCOMES:
Skin reactions according to Holgers | At time of sugical follow up visit (visit window of 7-14 days after surgery)
  Focus is on healing, post-operative complications and skin reactions after the first 7-14 days after surgery.

SECONDARY OUTCOMES:
Fitting of sound processor at surgical follow-up visit | At time of surgical follow up visit (visit window of 7-14 days after surgery)
  Implant stability is monitored before and after sound processor fitting through ISQ and clinical assessments.

OTHER OUTCOMES:
Surgical time | Recorded at surgery visit
  Time taken to perform the surgery
Surgical complications | At the surgical visit
  Any complications during and after surgery
Surgical complications | At time of surgical follow up visit (visit window of 7-14 days after surgery)
  Any complications during and after surgery
Implant stability | Duration of study (12 months of enrollment)
Use of Healing cap II | At the surgical visit
  Ease of use of Healing cap II and effect on surgical dressing
Use of Healing cap II | At time of surgical follow up visit (visit window of 7-14 days after surgery)
  Ease of use of Healing cap II and effect on surgical dressing
Skin healing at first follow-up visit | At time of surgical follow up visit (visit window of 7-14 days after surgery)
Pain and numbness | Duration of study (12 months of enrollment)
Time of fitting and type of sound processor | Duration of study (12 months of enrollment)

CONTACTS AND LOCATIONS:
Overall Officials: Søren Foghsgaard, M.D., Principal Investigator — Soeren.Foghsgaard@regionh.dk
Locations (2):
- Denmark (2):
  - Dept. of Otolaryngology - Head & Neck Surgery and Audiology, Gentofte/Rigshospitalet, Gentofte Municipality, Hellerup
  - Department of Oto-Rhino-Laryngology & Audiology, Aalborg University Hospital, Aalborg

IPD SHARING:
Plan to Share IPD: No